CLINICAL TRIAL: NCT01212016
Title: Immunopathogenesis of Food Allergy and Eosinophilic Gastrointestinal Disorders
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100196; 10-I-0196
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2015-05-13

CONDITIONS: Eosinophilic Gastroenteritis; Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; Eosinophilic Gastroenteritis; Peanut Allergy; T Cell; IgE; Food Allergy
MeSH Terms: conditions — Eosinophilic enteropathy; Eosinophilic Esophagitis; Peanut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Food allergies are characterized by abnormal immune system responses to certain foods, such as peanuts, strawberries, and shellfish. Some individuals with these allergies have immediate allergic reactions on contact with the food in question and need immediate treatment to prevent severe complications. In contrast, eosinophil-associated gastrointestinal disorders are related disorders in which white blood cells in the intestinal tract react to certain foods, causing abdominal pain, nausea, and other digestion problems. Researchers are interested in studying these conditions to better understand how the immune system responds to food allergies.

Objectives:

* To examine how the immune system responds to food allergens.
* To examine how certain white blood cells contribute to disease in individuals with food allergies and other inflammatory diseases.

Eligibility:

* Individuals between 18 and 65 years of age who have a history of (a) severe allergic reaction to peanuts (and have peanut-specific antibodies), (b) allergy or inflammatory disease, or (c) eosinophil-associated gastrointestinal disorder (with at least two documented food allergies).
* Healthy volunteers between 18 and 65 years of age who have no known allergies or asthma.

Design:

* All participants will have a screening visit and a procedure visit. The procedure visit will take place within 30 to 60 days of the screening visit, and will take 3 to 4 hours depending on the procedure(s) done.
* Participants will be screened with a physical examination and medical history, and will provide blood samples for testing. Participants with peanut or other allergies will have additional tests to determine their levels of sensitivity to certain foods. Participants with eosinophil-associated gastrointestinal disorder will provide stool samples for testing.
* At the procedure visit, participants with peanut allergies and participants with other allergies will provide blood samples and have leukapherisis to collect white blood cells for examination.
* At the procedure visit, healthy volunteers and participants with eosinophil-associated gastrointestinal disorder will provide blood samples and have leukapherisis to collect white blood cells for examination. In addition, some but not all of these participants will have a procedure called esophagogastroduodenoscopy (EGD), which will examine the esophagus, stomach, and small intestine. Participants who are scheduled to have EGD will be asked to fast for 6 hours before the procedure.

DETAILED DESCRIPTION:
Food allergy refers to a number of disorders characterized by clinical diseases associated with abnormal immune responses to food antigens. Classical IgE mediated anaphylactic food allergy is characterized by immediate hypersensitivity, and has a prevalence of approximately 6% and 3% in children and adults, respectively. In contrast, eosinophil associated gastrointestinal disorders (EGIDs), including eosinophilic esophagitis (EoE) and eosinophilic gastroenteritis (EG), are food allergy associated disorders characterized by eosinophilic inflammation of the gut, typically without anaphylaxis. Progress in the treatment and management of these food allergies requires further understanding of the immunological pathogenesis of these disorders. A subset of peripheral blood food allergen specific interleukin (IL) -5 producing T cells that are present in EGID but not peanut allergic subjects has recently been characterized. The primary objective of this study is to determine if similar IL-5 producing T cells are present in the gut of EGID subjects. To this end, both EGID and healthy non-allergic subjects will be enrolled and gastrointestinal biopsies will be obtained for intracellular cytokine staining, RT-PCR and ELISA.

Additionally, this protocol will supply blood and leukapheresis samples for exploratory studies on immunologic mechanisms underlying anaphylactic food allergy and EGIDs. A total of up to 400 subjects recruited from outside physician referrals and support groups, as well as from those in existing National Institutes of Health (NIH) protocols will be enrolled in this Clinical Center study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must meet all of the inclusion criteria:

All Subjects must:

1. Be willing to have samples collected and stored for future research.
2. Have a documented clinical history compatible with EGID, peanut allergy, or other allergic and inflammatory diseases or be healthy without known allergic conditions.

In addition to the above inclusion criteria for all subjects, the subjects in the following groups must meet additional group-specific inclusion criteria.

Subjects with EGID must:

1. Be greater than or equal to 18 years of age
2. Maintain a primary non-NIH physician for routine care
3. Have one of the types of EGID below:

   * Eosinophilic gastroenteritis: Have a clinical history of eosinophilic gastroenteritis -including gastrointestinal symptoms-, and histological evidence of stomach or duodenal eosinophilia with no other known etiology for the eosinophilia despite careful clinical evaluation.

OR

-Eosinophilic esophagitis: Have a diagnosis of eosinophilic esophagitis, including evidence of esophageal dysfunction with a peak count of greater than or equal to 25 eosinophils per high powered field, for which the biopsy was obtained while under proton pump inhibitor treatment.

OR

-Probable eosinophilic esophagitis: Have a likely diagnosis of eosinophilic esophagitis, based on evidence of esophageal dysfunction and a peak count of greater than or equal to 15 eosinophils per high powered field, but for which the biopsy was not obtained under proton pump inhibitors (per section 6.3). To confirm

a diagnosis of EoE, these subjects may be treated with proton pump inhibitor therapy at recommended doses for gastroesophageal reflux disease for at least 84 weeks prior to EGD and biopsy. The decision to recommend diagnostic biopsy will be according to concensus guidelines [7] and current standards of care: based on the severity of symptoms, history of food impactions, and evidence of remodeling (strictures).

Subjects with Peanut Allergy:

1. Be greater than or equal to 18 years of age and less than or equal to 65 years of age.
2. Have a history of immediate hypersensitivity to peanuts with involvement of at least one extracutaneous site, including wheezing, laryngeal edema, angioedema, vomiting, diarrhea, hypotension and circulatory collapse.
3. Have peanut specific IgE of greater than or equal to 5 kIU/L.

Subjects with Other Allergic and Inflammatory Diseases:

1. Be greater than or equal to 18 years of age and less than or equal to 65 years of age.
2. These subjects must be diagnosed with an allergic or an inflammatory disease, including anaphylaxis, asthma, or hay fever. Diagnosis will be based on established criteria for each clinical entity.

Healthy, Non-Atopic Subjects:

1. Be greater than or equal to 18 years of age and less than or equal to 65 years of age.
2. Have no history of allergies, asthma or food allergy
3. Have a negative ImmunoCAP fx5 in vitro food allergy screen for allergen specific IgE to egg white, milk, cod, wheat, peanut, and soy
4. Have a negative Phadiatop allergy screen

EXCLUSION CRITERIA:

Subjects with any of the following criteria will be excluded:

1. Any other condition that, in the investigator s opinion, places the subject at undue risk by participating in the study

Subjects with Peanut Allergy with any of the following will be excluded:

1. Chronic upper GI symptoms that are consistent with EGID (dysphagia, nausea, vomiting, abdominal pain/cramps, early satiety)

PROCEDURAL INCLUSIONS:

Subjects with EoE and EG undergoing research EGD or lymphapheresis must:

1. Be greater than or equal to 18 years of age and less than or equal to 65 years of age.

Subjects with EG undergoing EGD or lymphapheresis must have:

1. Histological evidence of stomach or duodenal eosinophilia with a peak count greater than or equal to 40 eosinophils per high powered field
2. Greater than two positive allergen skin tests or antigen specific IgE tests out of the following panel (peanut, wheat, soy, shrimp, egg white, milk, walnut, cod, corn)

Subjects with either EG or EoE undergoing lymphapheresis must have:

1. An absolute eosinophil count of >750 eos/microL at least once in the last 2 years

Subjects with EoE undergoing EGD must have:

1. Diagnosed EoE per section 5.1 with a previous biopsy showing greater than or equal to 25 eosinophils per high powered field, OR
2. Probable eosinophilic esophagitis per section 5.1 with a previous biopsy showing greater than or equal to 25 eosinophils per high powered field

PROCEDURAL EXCLUSIONS:

Subjects with any of following will not undergo EGD:

1. Uncontrolled asthma or Grade 3 or higher by the American Society of Anesthesiologist s (ASA) Physical Status Classification System.
2. History of adverse reaction to conscious sedation required for EGD.

Subjects with any of following will not undergo EGD or lymphapheresis:

1. Hemoglobin <12 g/dL
2. Viral screens positive for HIV or hepatitis B or C
3. Pregnant or breast-feeding women

Control Subjects (Healthy, Non-Atopic) Undergoing EGD with any of the following will be excluded:

1. History of reflux or use of acid suppression medication within the last 6 months.
2. Chronic gastrointestinal disease or immunological disease.
3. Clinically indicated EGD in the past 12 months.
4. Use of systemic corticosteroids in the past 6 months.

EGID subjects who are pregnant or breast-feeding may be followed without research phlebotomy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2010-08-30; Study Completion 2015-05-13

PRIMARY OUTCOMES:
Quantitation of gut tissue IL-5+ and IL-5- Th2 cells in EGIDs and in healthy non-atopic subjects. | End of study
Quantitation of gut tissue Th2 cells using alternative techniques (GATA3 immunohistochemistry, RT-PCR) in EGIDs and in healthy non-atopic subjects. | End of study
Quantitation of gut tissue IFN-, IL- 17 and IL-10 producing cellpopulations in EGIDs and in healthy non-atopic subjects. | End of study

SECONDARY OUTCOMES:
Characterization of gut homing food allergen specific T cells | End of study
Characterization of Pro-anaphylactic follicular helper Th2 cells in foodallergy | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Calman P Prussin, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Furuta GT, Liacouras CA, Collins MH, Gupta SK, Justinich C, Putnam PE, Bonis P, Hassall E, Straumann A, Rothenberg ME; First International Gastrointestinal Eosinophil Research Symposium (FIGERS) Subcommittees. Eosinophilic esophagitis in children and adults: a systematic review and consensus recommendations for diagnosis and treatment. Gastroenterology. 2007 Oct;133(4):1342-63. doi: 10.1053/j.gastro.2007.08.017. Epub 2007 Aug 8. PMID 17919504
- [Background] Sicherer SH, Sampson HA. Food allergy: recent advances in pathophysiology and treatment. Annu Rev Med. 2009;60:261-77. doi: 10.1146/annurev.med.60.042407.205711. PMID 18729729
- [Background] Sampson HA, Munoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, Brown SG, Camargo CA Jr, Cydulka R, Galli SJ, Gidudu J, Gruchalla RS, Harlor AD Jr, Hepner DL, Lewis LM, Lieberman PL, Metcalfe DD, O'Connor R, Muraro A, Rudman A, Schmitt C, Scherrer D, Simons FE, Thomas S, Wood JP, Decker WW. Second symposium on the definition and management of anaphylaxis: summary report--Second National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network symposium. J Allergy Clin Immunol. 2006 Feb;117(2):391-7. doi: 10.1016/j.jaci.2005.12.1303. PMID 16461139
- [Derived] Wansley DL, Yin Y, Prussin C. The retinoic acid receptor-alpha modulators ATRA and Ro415253 reciprocally regulate human IL-5+ Th2 cell proliferation and cytokine expression. Clin Mol Allergy. 2013 Dec 6;11(1):4. doi: 10.1186/1476-7961-11-4. PMID 24314292